CLINICAL TRIAL: NCT06342726
Title: The Effect of Active External Rewarming on Rewarming Rate in Simulated Prehospital Accidental Hypothermia - an Experimental Field Study
Brief Title: The Effect of Active External Rewarming on Rewarming Rate in Simulated Prehospital Accidental Hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024/714469
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Accidental Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Intervention Model Description: The study will use a crossover design on where research participants will undergo repetitions of the same scenario with different interventions in order to serve as their own control. The research participants will be healthy volunteers providing both oral and written consent.
  Before the start of experiment, the research participant will be cooled in an ice cave wearing wet clothing and with 2-3 m/s wind to a core temperature of 35.0 °C using the established protocol for inhibition of shivering. The maximum cooling time will be 2 hours (120 minutes). The order of interventions will be randomized.
  When the research subjects reach the target temperature of 35.0°C or the maximum cooling time of 2 hours, they will be subjected to one of the two scenarios listed below, with a rewarming phase of maximum 60 minutes.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Passive rewarming (Placebo Comparator): Wrapping of participants using a 3-layered model with a vapor barrier, insulating materials and an outer shell.
  Interventions: Device: Passive insulation
- Active rewarming (Active Comparator): Same as "Passive rewarming" but with an added external heat source
  Interventions: Device: PAX Warming Blanket; Device: Passive insulation

INTERVENTIONS:
Device: PAX Warming Blanket — Electric resistive active external warming blanket
  Arms: Active rewarming
Device: Passive insulation — 3-layered wrapping model

SUMMARY:
In this study, we aim to compare the effect of active external rewarming to passive rewarming in healthy research participants on core temperature.

The participants will be cooled to a core temperature of 35 degress C, the rewarmed using 2 different scenarios. Scenario 1 will be with passive rewarming, scenario 2 with active rewarming. Shivering will be pharmacologically inhibited using Buspirone and Meperidine.

DETAILED DESCRIPTION:
Accidental hypothermia is defined as an involuntary drop in core body temperature below 35°C. Hypothermia is a risk factor for cardiac arrythmia, pulmonary oedema, coagulopathy and neurological pathology. Isolated accidental hypothermia is potentially lethal on its own, and it is also an independent risk factor for increased mortality in patients with traumatic injury.

When core temperature drops, the body will automatically activate compensatory mechanisms in order to both increase thermic production and minimize heat loss in order to restore normal temperature. The mechanisms for thermal homeostasis are complex, strictly regulated and effective.

Until quite recently, active external rewarming was considered to be harmful and dangerous for patients with accidental hypothermia. A fear of fatal complications such as increased afterdrop and "rearming syndrome" leading to dangerous arrythmias and a drop in blood pressure which in a worst case scenario could lead to circulatory collapse, shock and potentially death.

Given the potentially detrimental consequences of being cold, any advice to abstain from warming patients should be well-documented, and the adverse effects of warming should outweigh those of being hypothermic. The lack of evidence for this claim that active external rewarming is dangerous along with many reports of successful external rewarming is leading to a change in most guidelines where active external rewarming is now an advisable treatment option.

A variety of different technological devices exist for the purpose of rewarming, but there is no established standard which is proven superior to others. Several trials have compared different rewarming methods, but evidence is limited. There is particularly deficient evidence regarding the amount of heat available for transfer from different methods and also the required amount of heat transfer for the rewarming to have a significant clinical impact.

Given the relatively short time in which active external rewarming has been advised, we suspect there is still a huge amount of room for improvement of care and technological innovation.

There is however reason to be cautious with active external rewarming of hypothermic patients. In a normothermic patient with normal circulatory function, thermal energy will be absorbed by the blood which flows back into central circulation distributing the heat evenly into a large volume. In a hypothermic patient there will be less cutaneous blood flow and less heat will be transferred to systemic circulation. This means that heat will accumulate on the skin surface and increase the risk of cutaneous injury, and there are several reported cases of this.

Hypothermia research with volunteer research participants is a complicated matter for many reasons. One complicating factor is shivering, which is an autonomic defense mechanism in which the muscles contract rapidly producing heat. It is the most effective method for the body to increase the metabolic heat production and re-establish normothermia. The shivering response is complicated in a research setting because there is a large interindividual variation in temperature threshold for initiation of shivering and in shivering intensity. This means that if you cool research participants down they will start to shiver at different core temperatures and with different intensities. Standardization of data is therefore impossible, and the researcher will be measuring the interindividual shivering abilities of the different research participants instead of the effect of the intervention. Shivering must therefore be inhibited in order to achieve reliable data.

ELIGIBILITY:
Participants are eligible to be included in the study only if all of the following criteria apply:

Age

1. Participant must be over 18 and under 40 years of age at the time of signing the informed consent.

   Type of Participant and Disease Characteristics
2. Participants who are overtly healthy as determined by their medical history. The participants will be asked to fill out a health-report stating to be healthy, using no relevant medication, and having no relevant allergies or hypersensitivity to the active substances or to any of the excipients of the medications used.

   Weight
3. BMI under 30 kg/m2 Sex and Contraceptive/Barrier Requirements 4. Both male and female participants can be included. Female participants of childbearing potential will be asked to take a pregnancy test to confirm the absence of pregnancy prior to study drug administration on both visit 1 and 2.

Informed Consent 5. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria Ahead of trial the participants will be contacted by a medical physician in the research group who will go through a medical questionnaire mainly based on the SmPC of Meperidine, Buspirone and Sodium chloride in "Felleskatalogen" with the following exclusion criteria.

1. Drugs: Concomitant use of sedatives, MAO-inhibitors, SSRI, ritonavir, cimetidine, chlorpromazine, phenytoin, erythromycin, itraconazole, platelet inhibitors, Apomorphine, alcohol (during the trial period) or other opioids or opioid antagonists (during the trial period). History of drug dependency.
2. Recent head injury (last. 12 months), known increased ICP, seizures or epilepsy
3. Other: Known reduced liver- or kidney function, reduced respiratory drive, known supraventricular tachycardia or prolonged QTc, hypertrophy of the prostate or urinary constriction, ongoing pregnancy or breastfeeding. Known acute glaucoma, myasthenia gravis. Previous abdominal surgery. History of cold injuries or frostbites.
4. Planned MRI the next two days after ingestion of temperature capsule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
Core body temperature | 2 hour cooling phase, 1 hour rewarming phase
  Esophageal measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mydske S, Helland AM, Borasio N, Brattebo G, Osteras O, Wiggen O, Assmus J, Strapazzon G, Thomassen O. Effect of active external rewarming on esophageal temperature in simulated prehospital accidental hypothermia: a randomized crossover trial. Scand J Trauma Resusc Emerg Med. 2025 Dec 12. doi: 10.1186/s13049-025-01528-7. Online ahead of print. PMID 41388306